CLINICAL TRIAL: NCT02690870
Title: Comparison of Tamoxifen and Clomiphene Citrate in Mild Stimulation IVF: a Prospective Cohort Study
Brief Title: Tamoxifen and Clomiphene Citrate in Mild Stimulation IVF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haiyan Lin, attending doctor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160220
Record Dates: First submitted 2016-02-20; First posted 2016-02-24 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
Keywords: tamoxifen; clomiphene; mild stimulation; poor ovarian response; clinical pregnancy rate
MeSH Terms: conditions — Infertility | interventions — Tamoxifen; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tamoxifen (Experimental): All patients will have serum hormone examination and be monitored by transvaginal ultrasound for ovaries on the day 3 of the menses（D3）.Patients in the tamoxifen group will take 20 mg of tamoxifen oral tablets daily from D3 for 5 days.All patients will check serum E2 and be monitored by transvaginal ultrasound for the mean follicular diameter and endometrial thickness on the day 8 of the cycle. The investigators will add HMG and GnRH-ant according to follicular diameter,E2 and LH. Human chorionic gonadotropin(hCG) (5000-10000 IU IM) will be given when one follicle measured at least 18 mm is found. IVF or ICSI will be performed 34-36 h after hCG administration. All patients will receive luteal phase support with progesterone 60 mg im qd for 2 weeks.
  Interventions: Drug: Tamoxifen
- clomiphene (Active Comparator): All patients will have serum hormone examination and be monitored by transvaginal ultrasound for ovaries on the day 3 of the menses（D3）.Patients in clomiphene group will take 100 mg of CC oral tablets daily from D3 for 5 days.All patients will have sexual hormone determination and be monitored by transvaginal ultrasound for the mean follicular diameter and endometrial thickness on the day 8 of the cycle.The investigators will add HMG and GnRH-ant according to follicular diameter,E2 and LH. Human chorionic gonadotropin(hCG) (5000-10000 IU IM) will be given when one follicle measured at least 18 mm is found. IVF or ICSI will be performed 34-36 h after hCG injection. All patients will receive luteal phase support with progesterone 60 mg im qd for 2 weeks.
  Interventions: Drug: Clomiphene

INTERVENTIONS:
Drug: Tamoxifen — Patients in the tamoxifen group will take 20 mg of tamoxifen oral tablets daily from day 3 of the menses for 5 days.
  Other Names: CAS RN：10540-29-1
  Arms: tamoxifen
Drug: Clomiphene — Patients in clomiphene group will take 100 mg of CC oral tablets daily from day 3 of the menses for 5 days.
  Other Names: clomiphene citrate
  Arms: clomiphene

SUMMARY:
The purpose of this prospective cohort study is to compare IVF outcome between tamoxifen and clomiphene citrate in mild stimulation.

DETAILED DESCRIPTION:
The reported prevalence of poor ovarian responders amongst patients undergoing IVF-ET is 9%-24%, and morbidity must be higher nowadays. For these women, Mild stimulation has been an important ovulation induction protocol. Clomiphene citrate(CC) and tamoxifen(TMX) are commonly used in mild stimulation protocol. It's reported that CC has adverse effect on growth of endrometrium and results in thin endrometrium(≤7mm) which maybe affect pregnancy rate. However, TMX has estrogen-like effect on the endrometrium that may be helpful to increase endormetrial thickness. The reported results about comparing CC with TMX showed that they had similar ovulation rate. Prospective study is necessary to confirm whether TMX is superior to CC on the IVF outcome.

ELIGIBILITY:
Inclusion Criteria:

1. age between 37 and 42;
2. BMI≤23kg/m2;
3. ≤3 oocytes with a conventional stimulation protocol;
4. AFC<5 follicles or AMH<1.1 ng/ml on the day 1 to 5 of the menses;
5. Cause of Infertiity: tubal factor, male factor, diminished ovarian reserve.

Exclusion Criteria:

1. endormetrial polyp, endormetrial cancer,intrauterine adhesions,uterine fibroids that affects uterine cavity
2. Endometriosis, adenomyosis
3. The diameter of Hydrosalpinx >2cm

Ages: 37 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-05 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | four weeks after embryo transfer

SECONDARY OUTCOMES:
cycle cancellations for thin endrometrial thickness | on the HCG day
endrometrial pattern and thickness on the day of HCG administration | on the HCG day
the number of follicular diameter≥10mm and sexual hormone test on the HCG day | on the HCG day

CONTACTS AND LOCATIONS:
Overall Officials: Qingxue ZHANG, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: Yes
Yes

REFERENCES:
- [Background] Boostanfar R, Jain JK, Mishell DR Jr, Paulson RJ. A prospective randomized trial comparing clomiphene citrate with tamoxifen citrate for ovulation induction. Fertil Steril. 2001 May;75(5):1024-6. doi: 10.1016/s0015-0282(01)01749-6. PMID 11334921
- [Background] Revelli A, Casano S, Salvagno F, Delle Piane L. Milder is better? Advantages and disadvantages of "mild" ovarian stimulation for human in vitro fertilization. Reprod Biol Endocrinol. 2011 Feb 16;9:25. doi: 10.1186/1477-7827-9-25. PMID 21324155
- [Background] Badawy A, Gibreal A. RETRACTED: Clomiphene citrate versus tamoxifen for ovulation induction in women with PCOS: a prospective randomized trial. Eur J Obstet Gynecol Reprod Biol. 2011 Nov;159(1):151-154. doi: 10.1016/j.ejogrb.2011.07.015. Epub 2011 Aug 9. No abstract available. PMID 21831503 (Retraction: PMID 35700607 Eur J Obstet Gynecol Reprod Biol. 2022 Aug;275:17)
- [Background] Wang CW, Horng SG, Chen CK, Wang HS, Huang HY, Lee CL, Soong YK. Ovulation induction with tamoxifen and alternate-day gonadotrophin in patients with thin endometrium. Reprod Biomed Online. 2008 Jul;17(1):20-6. doi: 10.1016/s1472-6483(10)60288-x. PMID 18616885
- [Background] Reynolds K, Khoury J, Sosnowski J, Thie J, Hofmann G. Comparison of the effect of tamoxifen on endometrial thickness in women with thin endometrium (<7mm) undergoing ovulation induction with clomiphene citrate. Fertil Steril. 2010 Apr;93(6):2091-3. doi: 10.1016/j.fertnstert.2009.08.038. Epub 2009 Sep 22. PMID 19775686
- [Background] Brinton LA, Westhoff CL, Scoccia B, Lamb EJ, Trabert B, Niwa S, Moghissi KS. Fertility drugs and endometrial cancer risk: results from an extended follow-up of a large infertility cohort. Hum Reprod. 2013 Oct;28(10):2813-21. doi: 10.1093/humrep/det323. Epub 2013 Aug 13. PMID 23943795
- [Background] Ozcan Cenksoy P, Ficicioglu C, Kizilkale O, Suhha Bostanci M, Bakacak M, Yesiladali M, Kaspar C. The comparision of effect of microdose GnRH-a flare-up, GnRH antagonist/aromatase inhibitor letrozole and GnRH antagonist/clomiphene citrate protocols on IVF outcomes in poor responder patients. Gynecol Endocrinol. 2014 Jul;30(7):485-9. doi: 10.3109/09513590.2014.893571. Epub 2014 Mar 5. PMID 24592985
- [Background] Pourmatroud E, Zargar M, Nikbakht R, Moramazi F. A new look at tamoxifen: co-administration with letrozole in intrauterine insemination cycles. Arch Gynecol Obstet. 2013 Feb;287(2):383-7. doi: 10.1007/s00404-012-2556-3. Epub 2012 Sep 25. PMID 23008110
- [Background] Mazzarino M, Biava M, de la Torre X, Fiacco I, Botre F. Characterization of the biotransformation pathways of clomiphene, tamoxifen and toremifene as assessed by LC-MS/(MS) following in vitro and excretion studies. Anal Bioanal Chem. 2013 Jun;405(16):5467-87. doi: 10.1007/s00216-013-6961-7. Epub 2013 Apr 23. PMID 23604525
- [Background] Brown J, Farquhar C, Beck J, Boothroyd C, Hughes E. Clomiphene and anti-oestrogens for ovulation induction in PCOS. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD002249. doi: 10.1002/14651858.CD002249.pub4. PMID 19821295
- [Background] Zakherah MS, Nasr A, El Saman AM, Shaaban OM, Shahin AY. Clomiphene citrate plus tamoxifen versus laparoscopic ovarian drilling in women with clomiphene-resistant polycystic ovary syndrome. Int J Gynaecol Obstet. 2010 Mar;108(3):240-3. doi: 10.1016/j.ijgo.2009.10.004. Epub 2009 Nov 26. PMID 19944418
- [Background] Steiner AZ, Terplan M, Paulson RJ. Comparison of tamoxifen and clomiphene citrate for ovulation induction: a meta-analysis. Hum Reprod. 2005 Jun;20(6):1511-5. doi: 10.1093/humrep/deh840. Epub 2005 Apr 21. PMID 15845599
- [Background] Wang HS, Wang TH, Soong YK. Cyclic changes in serum levels of insulin-like growth factor binding protein-1 in women treated with clomiphene citrate and tamoxifen. Gynecol Endocrinol. 2000 Aug;14(4):236-44. doi: 10.3109/09513590009167687. PMID 11075292
- [Background] Mazzarino M, Bragano MC, de la Torre X, Molaioni F, Botre F. Relevance of the selective oestrogen receptor modulators tamoxifen, toremifene and clomiphene in doping field: endogenous steroids urinary profile after multiple oral doses. Steroids. 2011 Nov;76(12):1400-6. doi: 10.1016/j.steroids.2011.06.005. Epub 2011 Jun 30. PMID 21745489